CLINICAL TRIAL: NCT01408212
Title: Effectiveness of Additional Acupuncture Therapy for Lung Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruiting
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Jun-Yong Choi, Associate professor, Korean Medicine Hospital of Pusan National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KCRC-IRB-2011009 & L-2011-170
Record Dates: First submitted 2011-07-28; First posted 2011-08-03 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Acupuncture Therapy

ARMS (1):
- Acupuncture therapy (Experimental)
  Interventions: Procedure: Acupuncture treatment

INTERVENTIONS:
Procedure: Acupuncture treatment — Acupuncture treatment will be performed by licensed doctors in Korean Medicine using 0.20 mm (diameter) X 0.30 mm (length) sized disposable acupuncture on seven to ten consecutive days after admission to the Korean Medicine Hospital of Pusan National University. At least two sessions and a maximum of five sessions of acupuncture therapy will be administered per day. Acupuncture points consist of common points and additional points selected for typical complaints common in patients under chemotherapy. These points are as follows.
  * Common points: LI4 (bilateral), LU5 (bilateral), LU7 (bilateral), BL13 (bilateral), BL23 (bilateral), SP3 (bilateral), LU9 (bilateral), ST36 (bilateral) and CV22
  * Additional points Nausea/vomiting PC6 (bilateral) Dyspepsia: CV12, LU6 (bilateral) Insomnia: Yintang, KI5 (bilateral) Pain: Ashi points (tender spots)

SUMMARY:
This study aims for evaluating the effectiveness, safety and feasibility of additional acupuncture therapy for lung cancer patients who are under chemotherapy in an inpatient setting. The acupuncture therapy will be administered during a resting period between cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Karnofsky Performance Status (KPS) 60% or more
* Undergoing antineoplastic chemotherapy for lung cancer
* Able to provide informed consent

Exclusion Criteria:

* Brain metastasis, stroke or major psychiatric diseases
* Active infection
* Severe heart disease
* Serious systemic diseases such as uncontrolled hypertension and diabetes mellitus
* Acupuncture therapy within the previous three months
* Communication disorder
* Unwillingness to participate in the trial
* Severe immunocompromised state (absolute neutrophils count < 1000/cubic mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change score of Functional Assessment of Cancer Therapy-Lung (FACT-L) scale from baseline | 7-10 days during a rest period between chemotherapy cycles

SECONDARY OUTCOMES:
Change score of Functional Assessment of Cancer Therapy-Lung (FACT-L) scale from baseline | 4-5 weeks from baseline (3-4 weeks after treatment termination)
Change score of Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT fatigue) Scale from baseline | Baseline, 7-10 days after baseline, 4-5 weeks after baseline
Change of general condition assessment using visual analogue scale from baseline | Baseline, 7-10 days after baseline, 4-5 weeks after baseline
Adverse events | From study enrollment to the last follow-up (a maximum of day 36)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Seong Kim, PhD, Principal Investigator — Pusan National University Yangsan Hospital; Jun-Yong Choi, MS, Principal Investigator — Korean Medicine Hospital of Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital and Korean Medicine Hospital of Pusan National University, Yangsan, Gyeongsangnam-do, South Korea